CLINICAL TRIAL: NCT04305847
Title: Satisfaction Assessment After Axillary Brachial Plexus Block for Distal Arm Surgery
Brief Title: Satisfaction Assessment After Axillary Block
Acronym: Qual'AXI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2020/480
Record Dates: First submitted 2020-02-20; First posted 2020-03-12 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Satisfaction, Patient
Keywords: Anaesthesia, regional; axillary brachial plexus block
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qual'AXI group: patients for whom distal arm surgery was performed under Axillary Brachial Plexus Block
  Interventions: Other: perioperative satisfaction assessment

INTERVENTIONS:
Other: perioperative satisfaction assessment — Satisfaction assessment at 24 and 48 hours post operatively by self-administered survey questionnaire based on different scales: Evan-LR, Net Promotor Score, Satisfaction score.

SUMMARY:
Satisfaction assessment at 24 and 48 hours post operatively, after Axillary Brachial Plexus Block for Distal Arm Surgery.

DETAILED DESCRIPTION:
Inclusion after distal Arm Surgery performed under Axillary Brachial Plexus Block.

Satisfaction assessment at 24 and 48 hours post operatively by self-administered survey questionnaire based on different scales: Evan-LR, Net Promotor Score, Satisfaction score.

ELIGIBILITY:
Inclusion Criteria:

* patients for whom distal arm surgery was performed under Axillary Brachial Plexus Block

Exclusion Criteria:

* Refusal, inability to consent
* inability to fill self-administered survey questionnaire
* pregnancy and breastfeeding
* surgery > 2 hours
* second surgical site requiring anaesthesia or analgesia
* chronic use of analgesia (including opioids) or illegal drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients for whom distal arm surgery was performed under Axillary Brachial Plexus Block in a single university hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Evan-LR score on day 2 | at 48 hours postoperative
  self administrated Evan-LR: "Evaluation du Vécu de l'Anesthésie LocoRégionale" 0-to-100 scale, with "100" indicating the best possible level of satisfaction and "0" the worst.

SECONDARY OUTCOMES:
Evan-LR score on day 1 | at 24 hours postoperative
  self administrated Evan-LR: "Evaluation du Vécu de l'Anesthésie LocoRégionale" 0-to-100 scale, with "100" indicating the best possible level of satisfaction and "0" the worst.
Net Promotor score on day 2 | at 48 hours postoperative
  self administrated Net Promotor score: willingness to advise a relative to undergo the same operation on a scale from 0 to 10. Based on the score, patients are divided into promoters (9 or 10), passives (7 or 8), and detractors (under 6). The NPS is determined as follows: NPS = % promoters - % detractors
Net Promotor score on day 1 | at 24 hours postoperative
  self administrated Net Promotor score: willingness to advise a relative to undergo the same operation on a scale from 0 to 10. Based on the score, patients are divided into promoters (9 or 10), passives (7 or 8), and detractors (under 6). The NPS is determined as follows: NPS = % promoters - % detractors
Patient Satisfaction score on day 2 | at 48 hours postoperative
  self administrated Satisfaction score: scale from 0 to 10. A score of "0" meant extremely dissatisfied and that a score of "10" meant extremely satisfied
Patient Satisfaction score on day 1 | at 24 hours postoperative
  self administrated Satisfaction score: scale from 0 to 10. A score of "0" meant extremely dissatisfied and that a score of "10" meant extremely satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) Sharing Statement depending on the institutional modality under development